CLINICAL TRIAL: NCT03224091
Title: PROspective Longitudinal All-comer Inclusion Study in Eating Disorders
Acronym: PROLED
Status: Recruiting | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Southern Denmark (Other); University of Copenhagen (Other); Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Jan Magnus Sjögren, Research Associate Professor, Sr Consultant Psychiatrist, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Other Study IDs: PCB-BCRED-1
Record Dates: First submitted 2017-03-23; First posted 2017-07-21 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Eating Disorder NOS
Keywords: Eating disorders; psychopathology; pathophysiology; prospective; longitudinal
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients at Psychiatric Center Ballerup
- Healthy Controls
- Healthy Controls recovered from an eating disorder

SUMMARY:
The PROLED study is a prospective and longitudinal study of patients with Eating Disorders. Annual interviews and collection of biological samples are done, as well as during changes in disease course e.g. during hospitalization. Included are qualitative interviews, psychometric tests, questionnaires which are used to collect data on psychopathology. There is also collection of blood, urine and faeces.

DETAILED DESCRIPTION:
The objective is to increase the understanding of the psychopathology and pathophysiology of Eating Disorders.

More specifically, the aim is to identify biomarkers that relate to prognosis, disease course and response to treatment as usual of Eating Disorders, and, to improve the understanding of the pathophysiology of Eating disorders in order to identify novel molecular targets for treatment.

Rationale The etiology of Eating Disorders (ED's) is unknown. Previous studies have identified genes that link Anorexia Nervosa to other psychiatric (e.g. schizophrenia) and somatic disorders (e.e. diabetes). Association studies have also suggested genetic causes underlying Bulimia Nervosa and Binge Eating Disorders. The PROLED study aims to improve the understanding of both the psychopathology and pathophysiology of Eating Disorders. No experimental drug will be used in this study.

There is a great need for an increased biological understanding of ED's in view of the prevalence, the costs, the severity and high mortality rates, and the lack of efficient treatments. The PROLED study aims to answer questions related to these unmet medical needs.

The study design is prospective and longitudinal. Qualitative interviews, psychometric tests, questionnaires are used to collect data on psychopathology. There is also collection of blood, urine and faeces.

ELIGIBILITY:
Inclusion Criteria:

* Eating Disorder (ICD-10)

Exclusion Criteria:

* Forced care/non-voluntary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at Psychiatric Center Ballerup with Eating Disorders
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-25 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
GAF-F total score | through study completion, an average of 1 year
  Change in Global level of functioning will be assessed using the GAF-F score for the whole population of treated individuals
BMI change over time | through study completion, an average of 1 year
  Change in Body Mass Index (BMI) will be assess in the whole population of Anorexia Nervosa patients and compared to other diagnoses and Healthy controls, change over time

SECONDARY OUTCOMES:
MDI | through study completion, an average of 1 year
  Change in Major Depressive Inventory will be used to assess depressiveness, assessed for all patients with one diagnosis and compared to other diagnoses and healthy controls; change over time
cytokines in plasma | through study completion, an average of 1 year
  Change in inflammatory parameters in blood as a measure of inflammation status
Biomarkers in blood | through study completion, an average of 1 year
  Change in biomarker parameters in blood as a measure of change in biological parameters
Total score on CogTrac | through study completion, an average of 1 year
  Change in cognitive performance
Change in EDI | through study completion, an average of 1 year
  Change in Eating disorder related behaviour and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Louise Behrend_Rasmussen, MD,PhD, Study Chair — Mental Health Center Ballerup
Locations (1):
- Mental Health Center, Ballerup Municipality, Capitol Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided